CLINICAL TRIAL: NCT05974696
Title: A Research Registry on Aggressive PitNETs
Acronym: RECAPitNETT
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0026
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Endocrine Tumor
Keywords: Endocrine Tumor; Reference centre; rare diseases; transcriptoms
MeSH Terms: conditions — Endocrine Gland Neoplasms; Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Anatomopathology samples collected and analysed as part of the routine care of the patient will be sent for centralised analysis to the Cochin Institute in Paris.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients RECAPitNETT: All adult subjects with pituitary tumours whose file is presented to the national HYPOcare RCP. There is only one group.

SUMMARY:
To allow the identification of markers, it is necessary to extend research networks more widely to collect and properly explore aggressive pituitary tumours. The multidisciplinary consultation meeting (RCP), organised by the reference centre for rare diseases of the pituitary gland, dedicated to aggressive pituitary tumours and carcinomas (HYPOcare), which is unique in France and brings together national experts, currently makes it possible to orientate the management of patients with an aggressive pituitary tumour. With more than 80 patient files discussed since its inception, the patient cohort via the HYPOcare RCP is one of the largest both nationally and internationally. At present, this data source is only dedicated to the clinical management of the files without the possibility of carrying out research work

ELIGIBILITY:
* Inclusion Criteria :

  * Patients with a diagnosis of pituitary tumour
  * Patients whose file has been presented to the national HYPOcare RCP
* Exclusion Criteria :

  * Patients objecting to participating in this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects with pituitary tumours whose file is presented to the national HYPOcare RCP. There is only one group.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2029-06-15 (Estimated); Study Completion 2029-06-15 (Estimated)

PRIMARY OUTCOMES:
Characterisation of aggressiveness of pituitary tumours by tanscriptome analysis | 3 years
  Molecular and transcriptomic signature of aggressiveness of pituitary tumours predictive of prognosis

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Groupement Hospitalier Est, Lyon, France